CLINICAL TRIAL: NCT02441491
Title: High-dose Cyclophosphamide for the Treatment of ROHHAD (Rapid Onset Obesity, Hypoventilation, Hypothalamic Dysfunction, and Autonomic Dysregulation) Syndrome
Brief Title: Treatment of Rapid Onset Obesity, Hypoventilation, Hypothalamic Dysfunction, and Autonomic Dysregulation (ROHHAD )
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate accrual
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00060912; J1520 (Other: SKCCC)
Record Dates: First submitted 2015-04-08; First posted 2015-05-12 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: ROHHAD Syndrome
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide (Experimental): Cyclophosphamide will be given by vein once a day for four straight days.
  Ten days after starting cyclophosphamide, filgrastim, a drug that helps normal blood cells to grow, will be given by vein once every day to try to help your blood cells grow faster.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide will be given by vein once a day for four straight days.
  Ten days after starting cyclophosphamide, filgrastim, a drug that helps normal blood cells to grow, by vein once every day to try to help your blood cells grow faster.
  Other Names: Cytoxan

SUMMARY:
ROHHAD (rapid onset obesity, hypothalamic dysfunction, hypoventilation, and autonomic dysregulation) syndrome is a rare pediatric disorder associated with a cancer called neuroblastoma and presumed to be driven by an attack of the immune system on specific area in the brain. Patients develop severe symptoms and often succumb to this disease. Based on the researchers' experience the investigators conduct a clinical trial to study intensive immunosuppression with high-dose cyclophosphamide in these patients. In addition to describing the symptomatic improvement, the investigators' trial seeks to define objective markers of disease activity.

DETAILED DESCRIPTION:
Baseline evaluation will include:

Sleep study and pulmonary evaluation Hormone levels Determination of up to 6 key ROHHAD-related symptoms to be followed Hyperphagia questionnaire 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) positron emission tomography (PET) scan Dual energy x-ray absorptiometry (DXA) scan Cerebrospinal fluid (CSF) analysis

Patients will be treated with cyclophosphamide, 50 mg/kg (ideal body weight)/dose daily for 4 days, with Mesna and hydration as prophylaxis against hemorrhagic cystitis. Supportive care will include mucosal care, transfusions, infection prophylaxis, and empiric treatment for febrile neutropenia.

Composite severity score will be assessed to measure response of key symptoms, and formal neuropsychological testing, sleep study, and hormone studies will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ROHHAD syndrome confirmed by two physicians.
* Any symptomatic improvement in response to a course of rituximab (five weekly doses) as assessed by parents and/or treating physician
* Normal brain MRI
* Cared for at home by the family
* Patients requiring bilevel positive airway pressure (BiPAP) support are eligible
* Negative pregnancy test for post pubertal female patients

Exclusion Criteria:

* Cardiac ejection fraction <40% or shortening fraction <20%.
* Inadequate pulmonary function, i.e. forced vital capacity or forced expiratory volume at one second < 50% of predicted for children greater than 8 years of age, or oxygen saturation <93% on pulse oximetry for younger children.
* Ventilator dependent
* Known chromosomal abnormality
* Active cancer diagnosis. Neuroblastoma that requires only follow up is eligible.
* Pregnancy

Ages: 12 Months to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Symptomatic improvement on the ROHHAD Symptoms Scale of children with ROHHAD syndrome after treatment with high-dose cyclophosphamide . | 18 months
Safety and toxicity of high-dose cyclophosphamide used to treat children with ROHHAD of as measured by NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0. | 18 months

SECONDARY OUTCOMES:
To calculate Area Under Curve (AUC) of high dose cyclophosphamide in obese children. | predose, 0, 1, 2, 4, 8, 12 and 24 hrs from the completion of infusion.
Neuropsychological function of patients with ROHHAD before and after high-dose cyclophosphamide measured using complementary age appropriate evaluation tools including Wechsler Preschool and Primary Scale of Intelligence RAN objects, and AIM. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Allen Chen, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Jacobson LA, Rane S, McReynolds LJ, Steppan DA, Chen AR, Paz-Priel I. Improved Behavior and Neuropsychological Function in Children With ROHHAD After High-Dose Cyclophosphamide. Pediatrics. 2016 Jul;138(1):e20151080. doi: 10.1542/peds.2015-1080. Epub 2016 Jun 16. PMID 27313069